CLINICAL TRIAL: NCT03191500
Title: Evaluate the Safety and Efficacy of a Steerable Catheter in the Treatment of Vascular Interventional Access : a Prospective, Muti-center, Single-arm Study
Brief Title: Evaluate the Safety and Efficacy of a Steerable Catheter in the Treatment of Vascular Interventional Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Wei Qiang Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT002
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- steerable catheter (Experimental): to study the safety and efficacy of a steerable catheter in the treatment of peripheral vascular disease
  Interventions: Device: steerable catheter

INTERVENTIONS:
Device: steerable catheter — peripheral vascular disease

SUMMARY:
This is a prospective, multicenter, single-arm clinical trial to evaluate safety and efficacy of a steerable catheter in the establishment of vascular intervention access. five centers participate in this study. The total enrollment number is 68. In the procedure of vascular interventional surgery or angiography diagnosis, the steerable catheter are used to building vascular interventional access. Evaluate the safety and efficacy of the product, by the observation and record the relative index of subjects intraoperative and postoperative (discharge) before and after 30 days .

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm clinical trial to evaluate safety and efficacy of a steerable catheter in the establishment of vascular intervention access. five centers participate in this study. The total enrollment number is 68. In the procedure of vascular interventional surgery or angiography diagnosis, the steerable catheter are used to building vascular interventional access. Evaluate the safety and efficacy of the product, by the observation and record the relative index(like catheter compliance, catheter directivity, and catheter visibility under X ray) of subjects in the procedure, telephone follow up at 30 days investigate the subjects healthy condition.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 80, male or female.
* Complying with the standard of peripheral vascular interventional operation treatment , complying with the standard treatment of vascular angiogram, need to establish vascular interventional treatment access.
* The subject who is able to understand the test purpose, voluntarily join this clinical trial with informed consent forms.

Exclusion Criteria:

* Patients with cerebrovascular accident or major gastrointestinal bleeding in six months unable to carry out antithrombotic therapy because of having contraindications to antiplatelet agents and anticoagulants and have haemorrhage tendency
* Hypohepatia, hematuria, deep vein thrombosis, and/or receiving the immunosuppressant therapy
* The distal target vessel blood flow low may produce thrombosis
* The women who pregnancy, lactation and can't contraception during the trial period
* Patients has been involved in other drugs or medical devices clinical trials related to treatment of the target lesion or has been involved in other drugs or medical device clinical trials but have not reached the primary endpoint of the study
* Patients unable or unwilling to participate in this trial
* the researcher determine the patient is not suitable to participate in clinical research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
procedure success rate | during the procedure
  The procedure success rate should fulfill the following three point at the same time:1 the steerable catheter can assist the guiding wire into the target vascular. 2 the steerable catheter can follow the guiding wire into the target vascular. 3 the steerable catheter can remove from the subject successfully.

SECONDARY OUTCOMES:
the steerable catheter compliance during the procedure of catheter access into the target vascular | during the procedure
  evaluate with excellent, good , general, poor four levels (according to surgeons experience to score)
the steerable catheter directivity during the procedure of catheter access into the target vascular | during the procedure
  evaluate with excellent, good , general, poor four levels (according to surgeons experience to score)
the steerable catheter visibility under the X-ray during the procedure of catheter access into the target vascular | during the procedure
  evaluate with excellent, good , general, poor four levels (according to surgeons experience to score)

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Fu, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No